CLINICAL TRIAL: NCT03418675
Title: A Double-Blind, Placebo-Controlled Study of Brexpiprazole in the Treatment of Borderline Personality Disorder.
Brief Title: Brexpiprazole in Borderline Personality Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-1729
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Results first posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 1 milligram per day for the first week and 1 milligram per day for the final taper week 2 milligrams per day for 10 weeks between taper periods.
  Interventions: Drug: Placebo
- Rexulti (Experimental): 1 milligram per day day for the first week and 1 milligram per day for the final taper week 2 milligrams per day for 10 weeks between taper periods.
  Interventions: Drug: Rexulti

INTERVENTIONS:
Drug: Rexulti — Atypical antipsychotic
  Other Names: Brexpiprazole
  Arms: Rexulti
Drug: Placebo — Pill that contains no medicine
  Other Names: no other names
  Arms: Placebo

SUMMARY:
The primary objective of the proposed study is to evaluate the safety and efficacy of Brexpiprazole in adults with borderline personality disorder (BPD). The hypothesis to be tested is that brexpiprazole will be more effective and well tolerated in adults with BPD compared to placebo. The proposed study will provide needed data on the treatment of a disabling disorder.

DETAILED DESCRIPTION:
Borderline personality disorder is characterized by mood instability, cognitive symptoms, impulsive behavior, and disturbed relationships (1-3). A variety of psychotherapies have been developed (4-6) and, while research on the use of medication is ongoing, no drug has been approved in the United States or elsewhere for its treatment (7). Second generation antipsychotics have been the most intensively studied (8-11). Current treatments for BPD are often inadequate. Dialectical behavioral therapy has been shown to reduce BPD but finding trained psychologists is difficult.

Dysfunctions in the serotoninergic and dopaminergic systems have been demonstrated in-and considered as possible causes for-symptoms associated with the disorder (25-28). Several studies on the use of traditional (29) and atypical antipsychotic agents in patients with borderline personality disorder (30-31) have shown a positive effect on individual symptoms (29, 32-36). However, we are not aware of any study evaluating Brexpiprazole in the treatment of patients with borderline personality disorder. In the proposed double-blind, placebo-controlled study, the influence of Brexpiprazole on the multifaceted psychopathological symptoms and aggression of patients with borderline personality disorder will be investigated.

Brexpiprazole therefore has distinctive properties that make it a promising option for patients with BPD. Brexpiprazole is a novel D2 partial agonist, has affinity for 5-HT1A, acts as an antagonist of the noradrenergic α1/2 receptor, partial agonist for D3, and antagonist for 5-HT2A (37-39). In addition, because of low rates of side effects, Brexpiprazole should be a well-tolerated and in fact desired medication approach to BPD.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 18-65;
2. Primary diagnosis of BPD
3. Zanarini scale score of at least 9 at baseline
4. Ability to understand and sign the consent form.

Exclusion Criteria:

1. Unstable medical illness based on history or clinically significant abnormalities on baseline physical examination
2. Subjects with schizophrenia or bipolar I disorder
3. Subjects with an active substance use disorder
4. Current pregnancy or lactation, or inadequate contraception in women of childbearing potential
5. Subjects considered an immediate suicide risk based on the Columbia Suicide Severity rating Scale (C-SSRS) (www.cssrs.columbia.edu/docs)
6. Illegal substance use based on urine toxicology screening
7. Initiation of psychological interventions within 3 months of screening
8. Use of any other psychotropic medication
9. Previous treatment with Brexpiprazole
10. Cognitive impairment that interferes with the capacity to understand and self-administer medication or provide written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, JD, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gunderson J: Borderline Personality Disorder, 2nd ed. Washington, DC, American Psychiatric Press, 2000
- [Background] Nakao K, Gunderson JG, Phillips KA, Tanaka N: Functional impairment in personality disorders. J Pers Disord 1992; 6:24-31
- [Background] Black DW, Blum N, Pfohl B, Hale N. Suicidal behavior in borderline personality disorder: prevalence, risk factors, prediction, and prevention. J Pers Disord. 2004 Jun;18(3):226-39. doi: 10.1521/pedi.18.3.226.35445. PMID 15237043
- [Background] Linehan MM, Comtois KA, Murray AM, Brown MZ, Gallop RJ, Heard HL, Korslund KE, Tutek DA, Reynolds SK, Lindenboim N. Two-year randomized controlled trial and follow-up of dialectical behavior therapy vs therapy by experts for suicidal behaviors and borderline personality disorder. Arch Gen Psychiatry. 2006 Jul;63(7):757-66. doi: 10.1001/archpsyc.63.7.757. PMID 16818865
- [Background] Blum N, St John D, Pfohl B, Stuart S, McCormick B, Allen J, Arndt S, Black DW. Systems Training for Emotional Predictability and Problem Solving (STEPPS) for outpatients with borderline personality disorder: a randomized controlled trial and 1-year follow-up. Am J Psychiatry. 2008 Apr;165(4):468-78. doi: 10.1176/appi.ajp.2007.07071079. Epub 2008 Feb 15. PMID 18281407
- [Background] McMain SF, Guimond T, Streiner DL, Cardish RJ, Links PS. Dialectical behavior therapy compared with general psychiatric management for borderline personality disorder: clinical outcomes and functioning over a 2-year follow-up. Am J Psychiatry. 2012 Jun;169(6):650-61. doi: 10.1176/appi.ajp.2012.11091416. PMID 22581157
- [Background] Lieb K, Vollm B, Rucker G, Timmer A, Stoffers JM. Pharmacotherapy for borderline personality disorder: Cochrane systematic review of randomised trials. Br J Psychiatry. 2010 Jan;196(1):4-12. doi: 10.1192/bjp.bp.108.062984. PMID 20044651
- [Background] Nickel MK, Muehlbacher M, Nickel C, Kettler C, Pedrosa Gil F, Bachler E, Buschmann W, Rother N, Fartacek R, Egger C, Anvar J, Rother WK, Loew TH, Kaplan P. Aripiprazole in the treatment of patients with borderline personality disorder: a double-blind, placebo-controlled study. Am J Psychiatry. 2006 May;163(5):833-8. doi: 10.1176/ajp.2006.163.5.833. PMID 16648324
- [Background] Schulz SC, Zanarini MC, Bateman A, Bohus M, Detke HC, Trzaskoma Q, Tanaka Y, Lin D, Deberdt W, Corya S. Olanzapine for the treatment of borderline personality disorder: variable dose 12-week randomised double-blind placebo-controlled study. Br J Psychiatry. 2008 Dec;193(6):485-92. doi: 10.1192/bjp.bp.107.037903. PMID 19043153
- [Background] Zanarini MC, Schulz SC, Detke HC, Tanaka Y, Zhao F, Lin D, Deberdt W, Kryzhanovskaya L, Corya S. A dose comparison of olanzapine for the treatment of borderline personality disorder: a 12-week randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2011 Oct;72(10):1353-62. doi: 10.4088/JCP.08m04138yel. PMID 21535995
- [Background] Pascual JC, Soler J, Puigdemont D, Perez-Egea R, Tiana T, Alvarez E, Perez V. Ziprasidone in the treatment of borderline personality disorder: a double-blind, placebo-controlled, randomized study. J Clin Psychiatry. 2008 Apr;69(4):603-8. doi: 10.4088/jcp.v69n0412. PMID 18251623
- [Background] Rinne T, de Kloet ER, Wouters L, Goekoop JG, de Rijk RH, van den Brink W. Fluvoxamine reduces responsiveness of HPA axis in adult female BPD patients with a history of sustained childhood abuse. Neuropsychopharmacology. 2003 Jan;28(1):126-32. doi: 10.1038/sj.npp.1300003. PMID 12496948
- [Background] Flewett T, Bradley P, Redvers A. Management of borderline personality disorder. Br J Psychiatry. 2003 Jul;183:78-9. doi: 10.1192/bjp.183.1.78-a. No abstract available. PMID 12835254
- [Background] Verheul R, Van Den Bosch LM, Koeter MW, De Ridder MA, Stijnen T, Van Den Brink W. Dialectical behaviour therapy for women with borderline personality disorder: 12-month, randomised clinical trial in The Netherlands. Br J Psychiatry. 2003 Feb;182:135-40. doi: 10.1192/bjp.182.2.135. PMID 12562741
- [Background] Nickel M, Nickel C, Leiberich P, Mitterlehner F, Forthuber P, Tritt K, Rother W, Loew T. [Psychosocial characteristics in persons who often change their psychotherapists]. Wien Med Wochenschr. 2004 Apr;154(7-8):163-9. doi: 10.1007/s10354-004-0058-z. German. PMID 15182043
- [Background] Nickel MK, Nickel C, Mitterlehner FO, Tritt K, Lahmann C, Leiberich PK, Rother WK, Loew TH. Topiramate treatment of aggression in female borderline personality disorder patients: a double-blind, placebo-controlled study. J Clin Psychiatry. 2004 Nov;65(11):1515-9. doi: 10.4088/jcp.v65n1112. PMID 15554765
- [Background] Nickel MK, Nickel C, Kaplan P, Lahmann C, Muhlbacher M, Tritt K, Krawczyk J, Leiberich PK, Rother WK, Loew TH. Treatment of aggression with topiramate in male borderline patients: a double-blind, placebo-controlled study. Biol Psychiatry. 2005 Mar 1;57(5):495-9. doi: 10.1016/j.biopsych.2004.11.044. PMID 15737664
- [Background] MacKinnon DF, Zandi PP, Gershon E, Nurnberger JI Jr, Reich T, DePaulo JR. Rapid switching of mood in families with multiple cases of bipolar disorder. Arch Gen Psychiatry. 2003 Sep;60(9):921-8. doi: 10.1001/archpsyc.60.9.921. PMID 12963674
- [Background] Crandell LE, Patrick MP, Hobson RP. 'Still-face' interactions between mothers with borderline personality disorder and their 2-month-old infants. Br J Psychiatry. 2003 Sep;183:239-47. doi: 10.1192/bjp.183.3.239. PMID 12948998
- [Background] Lieb K, Zanarini MC, Schmahl C, Linehan MM, Bohus M. Borderline personality disorder. Lancet. 2004 Jul 31-Aug 6;364(9432):453-61. doi: 10.1016/S0140-6736(04)16770-6. PMID 15288745
- [Background] Frankenburg FR, Zanarini MC. The association between borderline personality disorder and chronic medical illnesses, poor health-related lifestyle choices, and costly forms of health care utilization. J Clin Psychiatry. 2004 Dec;65(12):1660-5. doi: 10.4088/jcp.v65n1211. PMID 15641871
- [Background] Sher L, Oquendo MA, Li S, Huang YY, Grunebaum MF, Burke AK, Malone KM, Mann JJ. Lower CSF homovanillic acid levels in depressed patients with a history of alcoholism. Neuropsychopharmacology. 2003 Sep;28(9):1712-9. doi: 10.1038/sj.npp.1300231. Epub 2003 Jun 25. PMID 12825091
- [Background] Yen S, Shea MT, Sanislow CA, Grilo CM, Skodol AE, Gunderson JG, McGlashan TH, Zanarini MC, Morey LC. Borderline personality disorder criteria associated with prospectively observed suicidal behavior. Am J Psychiatry. 2004 Jul;161(7):1296-8. doi: 10.1176/appi.ajp.161.7.1296. PMID 15229066
- [Background] Zanarini MC, Frankenburg FR, Hennen J, Silk KR. The longitudinal course of borderline psychopathology: 6-year prospective follow-up of the phenomenology of borderline personality disorder. Am J Psychiatry. 2003 Feb;160(2):274-83. doi: 10.1176/appi.ajp.160.2.274. PMID 12562573
- [Background] Friedel RO. Dopamine dysfunction in borderline personality disorder: a hypothesis. Neuropsychopharmacology. 2004 Jun;29(6):1029-39. doi: 10.1038/sj.npp.1300424. PMID 15039763
- [Background] Hansenne M, Pitchot W, Pinto E, Reggers J, Scantamburlo G, Fuchs S, Pirard S, Ansseau M. 5-HT1A dysfunction in borderline personality disorder. Psychol Med. 2002 Jul;32(5):935-41. doi: 10.1017/s0033291702005445. PMID 12171388
- [Background] Nickel M, Leiberich P, Mitterlehner F: Atypical neuroleptics in personality disorders. Psychodynamic Psychotherapy 2003; 2:25-32
- [Background] Soloff PH, George A, Nathan S, Schulz PM, Cornelius JR, Herring J, Perel JM. Amitriptyline versus haloperidol in borderlines: final outcomes and predictors of response. J Clin Psychopharmacol. 1989 Aug;9(4):238-46. doi: 10.1097/00004714-198908000-00002. PMID 2768542
- [Background] Leucht S, Wahlbeck K, Hamann J, Kissling W. New generation antipsychotics versus low-potency conventional antipsychotics: a systematic review and meta-analysis. Lancet. 2003 May 10;361(9369):1581-9. doi: 10.1016/S0140-6736(03)13306-5. PMID 12747876
- [Background] Pascual JC, Oller S, Soler J, Barrachina J, Alvarez E, Perez V. Ziprasidone in the acute treatment of borderline personality disorder in psychiatric emergency services. J Clin Psychiatry. 2004 Sep;65(9):1281-2. doi: 10.4088/jcp.v65n0918b. No abstract available. PMID 15367057
- [Background] Zanarini MC, Frankenburg FR, Parachini EA. A preliminary, randomized trial of fluoxetine, olanzapine, and the olanzapine-fluoxetine combination in women with borderline personality disorder. J Clin Psychiatry. 2004 Jul;65(7):903-7. doi: 10.4088/jcp.v65n0704. PMID 15291677
- [Background] Ferreri MM, Loze JY, Rouillon F, Limosin F. Clozapine treatment of a borderline personality disorder with severe self-mutilating behaviours. Eur Psychiatry. 2004 May;19(3):177-8. doi: 10.1016/j.eurpsy.2003.11.004. No abstract available. PMID 15158928
- [Background] Bogenschutz MP, George Nurnberg H. Olanzapine versus placebo in the treatment of borderline personality disorder. J Clin Psychiatry. 2004 Jan;65(1):104-9. doi: 10.4088/jcp.v65n0118. PMID 14744178
- [Background] Zanarini MC, Frankenburg FR. Olanzapine treatment of female borderline personality disorder patients: a double-blind, placebo-controlled pilot study. J Clin Psychiatry. 2001 Nov;62(11):849-54. doi: 10.4088/jcp.v62n1103. PMID 11775043
- [Background] Zanarini MC. Update on pharmacotherapy of borderline personality disorder. Curr Psychiatry Rep. 2004 Feb;6(1):66-70. doi: 10.1007/s11920-004-0041-9. PMID 14738708
- [Background] Maeda K, Sugino H, Akazawa H, Amada N, Shimada J, Futamura T, Yamashita H, Ito N, McQuade RD, Mork A, Pehrson AL, Hentzer M, Nielsen V, Bundgaard C, Arnt J, Stensbol TB, Kikuchi T. Brexpiprazole I: in vitro and in vivo characterization of a novel serotonin-dopamine activity modulator. J Pharmacol Exp Ther. 2014 Sep;350(3):589-604. doi: 10.1124/jpet.114.213793. Epub 2014 Jun 19. PMID 24947465
- [Background] Maeda K, Lerdrup L, Sugino H, Akazawa H, Amada N, McQuade RD, Stensbol TB, Bundgaard C, Arnt J, Kikuchi T. Brexpiprazole II: antipsychotic-like and procognitive effects of a novel serotonin-dopamine activity modulator. J Pharmacol Exp Ther. 2014 Sep;350(3):605-14. doi: 10.1124/jpet.114.213819. Epub 2014 Jun 19. PMID 24947464
- [Background] Yoon S, Jeon SW, Ko YH, Patkar AA, Masand PS, Pae CU, Han C. Adjunctive Brexpiprazole as a Novel Effective Strategy for Treating Major Depressive Disorder: A Systematic Review and Meta-Analysis. J Clin Psychopharmacol. 2017 Feb;37(1):46-53. doi: 10.1097/JCP.0000000000000622. PMID 27941419
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Sheehan DV (1983). The Anxiety Disease. New York: Scribner's.
- [Background] Frisch MB, Cornell J, Villaneuva M (1993). Clinical validation of the Quality of Life Inventory: a measure of life satisfaction for use in treatment planning and outcome assessment. Psychol Assess. 4:92-101.
- [Background] Zanarini MC, Vujanovic AA, Parachini EA, Boulanger JL, Frankenburg FR, Hennen J. Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD): a continuous measure of DSM-IV borderline psychopathology. J Pers Disord. 2003 Jun;17(3):233-42. doi: 10.1521/pedi.17.3.233.22147. PMID 12839102
- [Background] Kay SR, Wolkenfeld F, Murrill LM. Profiles of aggression among psychiatric patients. I. Nature and prevalence. J Nerv Ment Dis. 1988 Sep;176(9):539-46. doi: 10.1097/00005053-198809000-00007. PMID 3418327
- [Background] Young RC, Biggs JT, Ziegler VE, Meyer DA. A rating scale for mania: reliability, validity and sensitivity. Br J Psychiatry. 1978 Nov;133:429-35. doi: 10.1192/bjp.133.5.429. PMID 728692
- [Background] Zanarini MC, Weingeroff JL, Frankenburg FR, Fitzmaurice GM. Development of the self-report version of the Zanarini Rating Scale for Borderline Personality Disorder. Personal Ment Health. 2015 Nov;9(4):243-9. doi: 10.1002/pmh.1302. Epub 2015 Jul 14. PMID 26174588
- [Background] Pfohl B, Blum N, St John D, McCormick B, Allen J, Black DW. Reliability and validity of the Borderline Evaluation of Severity Over Time (BEST): a self-rated scale to measure severity and change in persons with borderline personality disorder. J Pers Disord. 2009 Jun;23(3):281-93. doi: 10.1521/pedi.2009.23.3.281. PMID 19538082
- [Background] Barratt E: Anxiety and impulsiveness related to psychomotor efficiency. Percept Mot Skills 1959; 9:191-198
- [Background] Derogatis LR: SCL-90-R Administration, Scoring, and Procedures Manual II. Towson, Md, Clinical Psychometric Research, 1983
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Rexulti
Started | 40 | 40
Completed All Baseline Measures | 37 | 40
Completed One-post Randomization Visit | 34 | 35
Completed | 25 | 30
Not Completed | 15 | 10
Not completed — Lost to Follow-up | 13 | 10
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Population: Adults aged 18-65 years with a primary diagnosis of BPD and a Zanarini-BPD scale score of at least 9 at study entry who completed all baseline measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rexulti | Total
Number analyzed (Participants) | 37 | 40 | 77
Age, Continuous [Mean (Full Range); unit: years] | 28.9 [19 to 54] | 30.9 [19 to 61] | 29.9 [19 to 61]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 12 | 9 | 21
  Other | 4 | 2 | 6
  Unknown/Not reported | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 13 | 19 | 32
  Unknown or Not Reported | 16 | 14 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 7 | 13
  White | 22 | 20 | 42
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 6 | 9 | 15
Education [Count of Participants; unit: Participants]
  Less than HS diploma/GED | 0 | 0 | 0
  HS diploma/GED | 5 | 7 | 12
  Some college/Associates | 20 | 18 | 38
  Bachelors | 11 | 9 | 20
  Masters+ | 0 | 3 | 3
  Unknown/ Not Reported | 1 | 3 | 4
Employment Status [Count of Participants; unit: Participants]
  Full-time | 11 | 12 | 23
  Part-time | 2 | 3 | 5
  Student | 8 | 8 | 16
  Unemployed | 15 | 11 | 26
  Retired | 0 | 0 | 0
  Other | 1 | 1 | 2
  Unknown/Not Reported | 0 | 5 | 5
Marital Status [Count of Participants; unit: Participants]
  Single | 31 | 27 | 58
  Married | 2 | 3 | 5
  Divorced/separated | 3 | 6 | 9
  Living together/engaged | 1 | 1 | 2
  Widowed | 0 | 0 | 0
  Unknown/Not reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Zanarini Rating Scale for Borderline Personality Disorder
Description: A clinician-administered scale assessing Borderline Personality Scale severity at all study visits. Scores range from 0-36. Higher scores represent worse Borderline Personality Disorder severity, and lower scores represent milder Borderline Personality Disorder severity.
Time Frame: Baseline (Visit 1), Week 1 (Visit 2), Week 2 (Visit 3), Week 4 (Visit 4), Week 6 (Visit 5), Week 8 (Visit 6), Week 10 (Visit 7), Week 12 (Visit 8)
Population: Subjects assigned to Placebo or Rexulti who completed one-post randomization visit.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 34 | 35
score on a scale
  Visit 1 | 14.9 [9 to 26] | 14.9 [9 to 26]
  Visit 2 | 7.6 [0 to 19] | 6.7 [0 to 20]
  Visit 3 | 4.7 [0 to 16] | 5.3 [0 to 17]
  Visit 4 | 6 [0 to 18] | 4.4 [0 to 19]
  Visit 5 | 4.2 [0 to 15] | 4.5 [0 to 20]
  Visit 6 | 5.7 [0 to 14] | 4.9 [0 to 19]
  Visit 7 | 5 [0 to 16] | 4 [0 to 25]
  Visit 8 | 8.4 [0 to 22] | 3.1 [0 to 18]

2. Secondary Outcome: Modified Overt Aggression Scale (MOAS)
Description: A clinician-administered behavior rating scale measuring four types of aggressive behavior that will be assessed at all 9 visits. The subsets range on a scale from 0-4 with 0 indicating no aggression present. This scale tracks changes in level of aggression over time. The total weighted sum of the sections of the scale is recorded. Higher total scores indicate higher aggression levels.
Time Frame: as for outcome 1
Population: No data displayed because data were not collected. Due to the outbreak of the COVID-19 pandemic and following restrictions, all study visits were moved to teleheath and only essential scales were completed.
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Young Mania Rating Scale
Description: A clinician-administered, 11 item scale that assesses manic symptoms at baseline and over time. Higher total scores indicate higher severity of manic symptoms. This scale is used to rate the severity of manic abnormality in the patient. Subsets of the scale range from 0-4 with 0 indicating no severity. This scale will be assessed at all visits.
Time Frame: as for outcome 1
Population: as for outcome 2
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Self Report Version of Zanarini Scale
Description: A self-report scale assessing Borderline Personality severity that will be assessed at all visits.This scale is assessing severity and change in BPD symptoms. This is a 9-item scale measuring severity of different aspects of Borderline Personality Disorder, with each item rated on a 0-4 scale, 0=no symptoms, 4=severe symptoms. Total scores range from 0-36.
Time Frame: as for outcome 1
Population: Subjects assigned to Placebo or Rexulti who completed one-post randomization visit.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 34 | 35
score on a scale
  Visit 1 | 18.2 [8 to 36] | 17.6 [8 to 36]
  Visit 2 | 12.8 [0 to 36] | 10.9 [0 to 36]
  Visit 3 | 10.7 [0 to 36] | 7.9 [0 to 36]
  Visit 4 | 10.7 [0 to 36] | 8.0 [0 to 36]
  Visit 5 | 9.7 [0 to 36] | 7.0 [0 to 36]
  Visit 6 | 9.6 [0 to 36] | 6.6 [0 to 36]
  Visit 7 | 8.7 [0 to 36] | 6.0 [0 to 36]
  Visit 8 | 9.3 [0 to 36] | 5.8 [0 to 36]

5. Secondary Outcome: Borderline Evaluation of Severity Over Time (BEST)
Description: A self rated scale used to measure severity and change. The first 12 items of the scale are on a scale from 1-5, with 5 meaning that the item caused extreme distress, severe difficulties in relationships, and/or kept them from getting things done. The lowest rating (1) means it caused little or no problems. Items 13-15 (positive behaviors) are rated according to frequency. Completed at every visit.
Time Frame: Assessed at Visits 1 to 8, change in scores from Visit 1 to Visit 8 (baseline to week 12) is reported
Population: Subjects assigned to Placebo or Rexulti who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 25 | 30
score on a scale
  Visit 1 | 40.90 (10.91) | 40.54 (8.25)
  Visit 8 | 29.15 (8.37) | 23.15 (9.06)

6. Secondary Outcome: Barratt Impulsiveness Scale (BIS)
Description: A self-report assessment of impulsivity that will be assessed at baseline and visit 8. The BIS is composed of 30 items describing common impulsive or non-impulsive (for reverse scored items) behaviors and preferences. Items are scored on a 4-point scale: (Rarely/Never = 1, Occasionally = 2, Often = 3, Almost Always/Always = 4). These scores are summed to produce an overall impulsivity score ranging from 30 (not impulsive) to 120 (extremely impulsive).
Time Frame: Baseline (Visit 1), Week 12 (Visit 8)
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 25 | 30
score on a scale
  Visit 1 | 76.53 (15.33) | 72.27 (15.50)
  Visit 8 | 68.13 (13.89) | 70.5 (17.86)

7. Secondary Outcome: Symptom Checklist-90 Revised
Description: An instrument that helps evaluate a broad range of psychological problems and symptoms of Borderline Personality Disorder psychopathology. This will be assessed at baseline and visit 8.The 115 items are rated by using a 5-step Likert scale (0=not at all, 4=very strong) and provide a global picture of borderline psychopathology. Global scores of borderline psychopathology are calculated by summing 12 items and range from 0-48. Higher scores indicate more severe symptoms of Borderline Personality Disorder.
Time Frame: Baseline, Visit 8 (Week 12)
Population: Subjects who completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 25 | 30
score on a scale
  Visit 1 | 26.17 (10.44) | 25.42 (11.58)
  Visit 8 | 20.25 (7.99) | 14.21 (10.88)

8. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: A clinician-administered assessment of anxiety that will be assessed at all study visits (Visit 1-Visit 8). Changes in scores from baseline to final visit will be assessed. Higher scores (up to 56) indicate higher levels of anxiety, with 0 being no symptoms of anxiety.
Time Frame: assessed at Visits 1 to 8, change in scores from Visit 1 to Visit 8 (baseline to Week 12) is reported
Population: Subjects assigned to Placebo or Rexulti who completed the study.
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 25 | 30
change in score on a scale | -2.41 (8.43) | -4.88 (7.46)

9. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: A clinician-administered assessment of depression that will be assessed at all study visits (Visits 1-8). Higher total scores indicate higher levels of depression (up to 52), while a score of 0 would indicate no depressive symptoms.
Time Frame: Assessed at Visits 1 to 8, change in scores from Visit 1 to Visit 8 (baseline to week 12) is reported
Population: Subjects assigned to placebo or Rexulti who completed the study
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 25 | 30
change in score on a scale | -2.09 (6.91) | -3.81 (7.41)

10. Secondary Outcome: MINI International Neuropsychiatric Interview
Description: A short-structured interview that assesses comorbid psychiatric disorders according to the DSM 5 criteria. This assessment will be done during the baseline visit.
Time Frame: Baseline (Week 1)
Population: Subjects who completed all baseline measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 37 | 40
Participants
  Major Depressive Episode (Current) | 16 | 18
  Major Depressive Episode (Past) | 12 | 18
  Manic Episode (Current) | 2 | 2
  Manic Episode (Past) | 1 | 3
  Hypomanic Episode (Current) | 1 | 0
  Bipolar I Disorder (Current) | 0 | 0
  Bipolar I Disorder (Past) | 0 | 0
  Bipolar II Disorder (Current) | 0 | 0
  Bipolar II Disorder (Past) | 0 | 1
  Panic Disorder (Current) | 6 | 6
  Panic Disorder (Lifetime) | 11 | 10
  Agoraphobia (Current) | 7 | 9
  Social Anxiety Disorder (Current) | 6 | 9
  Obsessive Compulsive Disorder (Current) | 3 | 3
  Post Traumatic Stress Disorder (Current) | 9 | 12
  Alcohol Use Disorder (Past 12 months) | 13 | 8
  Substance Use Disorder (Past 12 months) | 11 | 8
  Any Psychotic Disorder (Current) | 0 | 0
  Any Psychotic Disorder (Lifetime) | 0 | 1
  Major Depressive Disorder with Psychotic Features (Current) | 0 | 0
  Major Depressive Disorder with Psychotic Features (Past) | 0 | 0
  Anorexia Nervosa (current) | 0 | 1
  Bulimia Nervosa (Current) | 4 | 4
  Binge Eating Disorder (Current) | 2 | 4
  Generalized Anxiety Disorder (Current) | 10 | 15
  Antisocial Personality Disorder (Lifetime) | 8 | 4
  ADHD Combined Type (Current) | 2 | 4
  ADHD Inattentive Type (Current) | 0 | 1
  ADHD Hyperactive Type (Current) | 1 | 1
  Tourette's Syndrome (Lifetime) | 0 | 1
  Persistent Motor Tic Disorder (Lifetime) | 1 | 1
  Provisional Vocal Tic Disorder (Lifetime) | 0 | 0
  Provisional Tic Disorder (Lifetime) | 0 | 0
  Specific Phobia | 4 | 1
  Body Dysmorphic Disorder (Current) | 3 | 2

11. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: Subjects will complete the SDS at all visits. The change in scores from baseline to study completion will be assessed. The scale itself assesses the level of disability from borderline personality disorder (or target disorder) with higher scores indicating a more debilitating disorder. Scores range from 0-30.
Time Frame: as for outcome 1
Population: Subjects who completed at least one post-randomization visit
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 34 | 35
score on a scale
  Visit 1 | 17.3 [0 to 30] | 15.8 [0 to 30]
  Visit 2 | 13.3 [0 to 30] | 10.7 [0 to 30]
  Visit 3 | 11.5 [0 to 30] | 7.8 [0 to 30]
  Visit 4 | 12.4 [0 to 30] | 7.8 [0 to 30]
  Visit 5 | 11.7 [0 to 30] | 7.0 [0 to 30]
  Visit 6 | 11.2 [0 to 30] | 7.9 [0 to 30]
  Visit 7 | 12.0 [0 to 30] | 6.9 [0 to 30]
  Visit 8 | 12.7 [0 to 30] | 7.7 [0 to 30]

12. Secondary Outcome: Quality of Life Inventory (QOLI)
Description: A self-report assessment of patient perceived quality of life that will be assessed at baseline and visit 8. Higher scores indicate a higher quality of life, whereas lower scores indicate a lower quality of life. Participants are asked to rate the importance of each domain on a 3-point scale ranging from 1=not important to 3=very important, and to rate how satisfied they are with that domain on a 6-point scale, ranging from -3=very dissatisfied to +3=very satisfied. In scoring, importance ratings are multiplied by satisfaction ratings to produce weighted satisfaction scores for each of the 16 domains. Weighted satisfaction scores are summed and divided by the number of domains that were rated as important or very important to produce a raw score, which is then converted to a t-score, which provides a proxy measurement for perceived quality of life. T-scores range from very low perceived quality of life (0-36) to high perceived quality of life (58-77).
Time Frame: Baseline (Week 1), Week 12 (Visit 8)
Population: Subjects who completed all visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 25 | 30
score on a scale
  Visit 1 | 28.89 (9.11) | 28.70 (11.18)
  Visit 8 | 30.75 (10.62) | 35.71 (6.43)

13. Secondary Outcome: Columbia Suicide Severity Rating Scale (CSSRS)
Description: A self-report scale measuring suicidality. Subjects will complete the scale at all visits. Subjects are asked about suicidal thoughts. If answers are no, rater can proceed to "suicidal behavior" section where subject is asked about any non-suicidal self injurious behavior. If yes, subject is asked about intensity of ideations. In the event of serious threat to themselves, the subject will be escorted to the emergency room. Total score indicates severity of suicidal ideation and behavior, with lower scores representing lower levels of suicidality and higher scores representing higher levels of suicidality. A score of 0 would reflect no suicidality present, whereas a maximum score of 5 would reflect active suicidal ideation with intent to act.
Time Frame: Baseline (Visit 1), Week 12 (Visit 8)
Population: Subjects who completed all baseline data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Rexulti
Number analyzed (Participants) | 40 | 40
score on a scale
  Visit 1 | 1.15 (1.72) | 0.73 (0.99)
  Visit 8 | 0.23 (0.66) | 0.08 (0.35)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 12 weeks.
Arm/Group | Placebo | Rexulti
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/40
Other Adverse Events (participants affected / at risk) | 19/40 | 11/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Rexulti (N=40)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) — Mild suicidal ideation without a plan. Serious as it necessitated hospitalization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | Rexulti (N=40)
Nausea (Gastrointestinal disorders) | 6 | 2
Fatigue (General disorders) | 4 | 2
Restlessness (General disorders) | 3 | 3
Dry Mouth (General disorders) | 0 | 3
Headache (General disorders) | 2 | 1
Hallucinations (Psychiatric disorders) | 2 | 0
Sleep Problems (General disorders) | 2 | 0
Tremor (General disorders) | 1 | 0
Sweating (General disorders) | 1 | 0
Increase Appetite (General disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT03418675/Prot_SAP_001.pdf